CLINICAL TRIAL: NCT01615874
Title: A Six-week Evaluator-Blind, Randomized, Active-Controlled Evaluation of the Effects of Three Doses of Mometasone Furoate/Formoterol Fumarate (MF/F) Metered Dose Inhaler (MDI), Montelukast, and Beclomethasone Dipropionate (BDP HFA) on the HPA Axis in Asthmatic Children 5 to 11 Years of Age (Protocol No. P05574/PN158)
Brief Title: Study of the Effect of Mometasone Furoate/Formoterol (MF/F), Montelukast and Beclomethasone Dipropionate (BDP) on Plasma Cortisol Levels of Children 5-11 Years Old With Persistent Asthma (P05574)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P05574; 2009-010108-27 (EudraCT Number)
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate, Formoterol Fumarate Drug Combination; Beclomethasone; montelukast; Aging; 3-(2-(4-azidobenzamidino)ethyl)-5-hydroxyindole; Prednisolone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- MF/F MDI 50/10 mcg BID (Experimental)
  Interventions: Drug: MF/F Metered Dose Inhaler (MDI) 25/5 mcg; Drug: Rescue medication: short-acting beta-2 agonist (SABA) MDI; Drug: Rescue medication: Prednisone/Prednisolone
- MF/F MDI 100/10 mcg BID (Experimental)
  Interventions: Drug: MF/F MDI 50/5 mcg; Drug: Rescue medication: short-acting beta-2 agonist (SABA) MDI; Drug: Rescue medication: Prednisone/Prednisolone
- MF/F MDI 200/10 mcg BID (Experimental)
  Interventions: Drug: MF/F MDI 100/5 mcg; Drug: Rescue medication: short-acting beta-2 agonist (SABA) MDI; Drug: Rescue medication: Prednisone/Prednisolone
- BDP HFA 160 mcg BID (Active Comparator)
  Interventions: Drug: BDP hydrofluoroalkane (HFA) 80 mcg; Drug: Rescue medication: short-acting beta-2 agonist (SABA) MDI; Drug: Rescue medication: Prednisone/Prednisolone
- Montelukast 5 mg QD (4 mg QD for 5-year-olds) (Active Comparator)
  Interventions: Drug: Montelukast tablets 5 mg (4 mg for children 5 years of age); Drug: Rescue medication: short-acting beta-2 agonist (SABA) MDI; Drug: Rescue medication: Prednisone/Prednisolone

INTERVENTIONS:
Drug: MF/F Metered Dose Inhaler (MDI) 25/5 mcg — MF/F MDI 25/5 mcg, 2 inhalations twice a day (BID)
  Other Names: SCH 418131; MK-0887A; DULERA®
  Arms: MF/F MDI 50/10 mcg BID
Drug: MF/F MDI 50/5 mcg — MF/F MDI 50/5 mcg, 2 inhalations BID
  Other Names: SCH 418131; MK-0887A; DULERA®
  Arms: MF/F MDI 100/10 mcg BID
Drug: MF/F MDI 100/5 mcg — MF/F MDI 100/5 mcg, 2 inhalations BID
  Other Names: SCH 418131; MK-0887A; DULERA®
  Arms: MF/F MDI 200/10 mcg BID
Drug: BDP hydrofluoroalkane (HFA) 80 mcg — BDP HFA 80 mcg, 2 inhalations BID
  Other Names: BECONASE AQ®; QVAR®
  Arms: BDP HFA 160 mcg BID
Drug: Montelukast tablets 5 mg (4 mg for children 5 years of age) — Montelukast chewable tablets 5 mg once daily (QD) for children 6-11 years of age
  OR
  Montelukast chewable tablets 4 mg QD for children 5 years of age
  Other Names: MK-0476; SINGULAIR®
  Arms: Montelukast 5 mg QD (4 mg QD for 5-year-olds)
Drug: Rescue medication: short-acting beta-2 agonist (SABA) MDI — albuterol MDI 90 mcg OR or salbutamol HFA MDI 100 mcg for rescue medication, taken as directed
Drug: Rescue medication: Prednisone/Prednisolone — Prednisone/Prednisolone for rescue medication, taken as directed

SUMMARY:
The purpose of this study is to assess the effect of one of five possible study medications used in the treatment of asthma on blood plasma cortisol levels in children aged 5-11 years with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of persistent asthma of ≥6 months duration
* body weight ≥18 kg
* able to discontinue prescribed inhaled corticosteroid (ICS) or ICS combined with long-acting beta-agonist (LABA) before starting study medication
* use of a low or medium daily dose of ICS (either alone or in combination with a LABA) with no use of oral corticosteroids within 3 months prior to Screening Visit
* stable asthma regimen (daily dose unchanged) for ≥2 weeks prior to Screening Visit
* documented positive responsiveness to bronchodilators
* ability to use a peak flow meter correctly and to perform spirometry and PEF measurements
* ability to use an inhaler correctly
* consent/assent for the trial and for pharmacogenetic testing (Note: If unwilling to consent/assent for pharmacogenetic testing, inclusion in the study is still allowed, but no pharmacogenetic samples will be obtained.)

Exclusion Criteria:

* use of a high dose of ICS for ≥30 days within 6 months prior to Screening Visit
* treatment in the emergency room (for a severe asthma exacerbation requiring systemic corticosteroid treatment) or hospitalization for management of airway obstruction within 3 months prior to Screening Visit
* ever required ventilator support for respiratory failure secondary to asthma
* upper or lower respiratory tract infection (viral or bacterial) within 2 weeks prior to Screening Visit
* clinically significant abnormal vital sign
* evidence of oropharyngeal candidiasis
* history of clinically significant renal, hepatic, cardiovascular, metabolic, neurologic, hematologic, ophthalmologic, respiratory, gastrointestinal, cerebrovascular, or other significant medical illness or disorder that may interfere with study participation. Specific examples include but are not limited to insulin-dependent diabetes, active hepatitis, cardiovascular disease including hypertension, or conditions that may interfere with respiratory function such as, bronchiectasis, and cystic fibrosis
* allergy to or intolerance of corticoids, beta-2 agonists, montelukast or any of the inactive ingredients in the medications used in this study
* participation in this same study at another study site
* previous randomization into this study
* participation in another investigational study for the duration of this study
* use of any investigational drug within one month prior to Screening Visit
* previous participation in a study with MF/F or montelukast
* direct association with or family member of one of the investigators or study staff
* sibling of a participant in this study

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Plasma Cortisol Area Under the Curve (AUC) 0-24 hrs | Baseline (Day 1) and Day 42

SECONDARY OUTCOMES:
Change from Baseline in Plasma Cortisol Trough Concentration (Ctrough) | Baseline (Day 1) and Day 42